CLINICAL TRIAL: NCT00580320
Title: Phase I Trial of Dacarbazine and Bortezomib in Melanoma and Soft Tissue Sarcoma
Brief Title: Safety Study of Dacarbazine and Bortezomib in Melanoma and Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-03740
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Melanoma; Soft Tissue Sarcoma; Parathyroid Carcinoma; Small Cell Carcinoma of the Lung; Carcinoid Tumors
Keywords: melanoma; soft tissue sarcoma; APUD tumor; dacarbazine; bortezomib; velcade
MeSH Terms: conditions — Melanoma; Sarcoma; Parathyroid Neoplasms; Small Cell Lung Carcinoma; Carcinoid Tumor | interventions — Dacarbazine; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): dacarbazine + bortezomib
  Interventions: Drug: Dacarbazine and bortezomib

INTERVENTIONS:
Drug: Dacarbazine and bortezomib — Level 0: Dacarbazine 190 mg/m2 + Bortezomib 1.0 mg/m2; Level 1: Dacarbazine 250 mg/m2 + Bortezomib 1.0 mg/m2; Level 2: Dacarbazine 250 mg/m2 + Bortezomib 1.3 mg/m2; Level 3: Dacarbazine 250 mg/m2 + Bortezomib 1.6 mg/m2; Level 4: Dacarbazine 330 mg/m2 + Bortezomib 1.6 mg/m2; Level 5: Dacarbazine 440 mg/m2 + Bortezomib 1.6 mg/m2; Level 6: Dacarbazine 580 mg/m2 + Bortezomib 1.6 mg/m2
  Other Names: bortezomib (velcade)

SUMMARY:
Bortezomib will enhance the activity of dacarbazine against melanoma and soft tissue sarcoma. Weekly administration of the combination will prove to be feasible and tolerable at an appropriate dose.

DETAILED DESCRIPTION:
The primary objective is to determine recommended phase II doses for the combination dacarbazine and bortezomib administered weekly.

Secondary objectives are to determine the maximum tolerated dose combination and to observe anti-tumor activity in terms of response rate(s), duration of response, time to progression, and time on treatment (a measure of both antitumor activity and treatment tolerance).

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of cutaneous or mucosal melanoma, soft tissue sarcoma (STS), or an APUD (amine precursor uptake and decarboxylation) tumor. APUD tumors include parathyroid carcinoma, medullary carcinoma of the thyroid, small cell carcinoma of the lung, pheochromocytoma, islet cell tumors, carcinoid tumors, and malignant paraganglioma.
* Measurable or evaluable disease not appropriate for resection and/or radiation with curative intent. Patients with small cell carcinoma must have extended stage disease or, if limited stage disease, must have received at least one prior systemic therapy.
* Age 18 years or greater
* ECOG Performance Status 0 or 1
* Women must be post-menopausal, infertile as the result of a surgical procedure, or willing to use a medically accepted form of birth control (abstinence, hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condon with spermicide) for the duration of study treatment. Men also must agree to use a medically accepted form of birth control for the duration of study treatment.

Exclusion Criteria:

* Uncontrolled brain metastatic disease
* Platelet count <100
* Absolute neutrophil count <1.5
* Blood transfusion or hematopoietic growth factors for cytopenia within one month of enrollment.
* Calculated or measured (Cockcroft and Gault formula) creatinine clearance <30 mL/minute
* AST > 3 times the upper limit of normal, unless elevation due to metastatic disease, in which case AST > 5 times the upper limit of normal
* Bilirubin > 2 mg/mL
* Grade 2 or greater peripheral neuropathy
* Hypersensitivity to bortezomib, boron, mannitol, or dacarbazine
* Pregnant or nursing
* Other investigational drugs within 14 days of enrollment
* Other medical or other condition(s) that in the opinion of the investigator/sub-investigator might compromise the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-09; Primary Completion 2009-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety as measured by serious adverse events | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Massey Cancer Center/Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- See also: Publication — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3618599/